CLINICAL TRIAL: NCT02219061
Title: Observation Study on Early Waning of Maternal Measles and Meningitis C Antibodies
Brief Title: Early Waning of Maternal Measles and Meningitis C Antibodies
Acronym: EWMM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Other Study IDs: GZCDC001
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-08

CONDITIONS: Measles
Keywords: Measles; Meningitis C; waning; Geometric Mean Titer; China
MeSH Terms: conditions — Measles

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Children's Serum will be collected for measles and meningitis C antibodies test by ELISA method.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GMT

SUMMARY:
Maternal antibodies (measles and meningitis C) may wane in the first six months after birth.

* Geometric mean titers(GMTs) of measles and meningitis C.
* Follow-up on 0 month, 3rd month,5th month and 7th month after birth.

DETAILED DESCRIPTION:
Measles and meningitis C are hot topics in China in recent years. Although China had set the goal of measles elimination, many measles cases were found to be those aged < 8 months and meningitis C is becoming public health issue since meningitis group A has been controlled at a very low level and little is known on C group. So the investigators designed the observation study on the two antibodies.

Maternal antibodies are supposed to wane after birth. Serums of the placenta(0 month), children of 3 months, 5 months and 7 months old will be collected and the geometric mean titers (GMTs) of measles and meningitis C will be confirmed by using the ELISA test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants.

Exclusion Criteria:

* Infants with poor score.

Max Age: 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer | Up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wang, Principal Investigator — Guangzhou CDC
Locations (1):
- Guangzhou Center for Disease Control and Prevention, Guangzhou, Guangdong, China